CLINICAL TRIAL: NCT01502618
Title: Development of a Secondary Prevention Intervention Targeting HIV-Positive Black Young Men Who Have Sex With Men
Brief Title: Intervention for HIV-Positive Black Young Men Who Have Sex With Men (YMSM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 090
Record Dates: First submitted 2011-03-10; First posted 2011-12-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-05

CONDITIONS: Acquired Immunodeficiency Syndrome
Keywords: Adolescent Medicine Trials Network for HIV/AIDS Interventions; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focus Group (Experimental): The focus group participants for this study will be Black Young Men who have Sex with Men (B-YMSM) ages 16-24 years (inclusive) who are diagnosed as HIV-positive and receive medical care at one of the two participating AMTUs or their community partners.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — N/A. Protocol is the focus group

SUMMARY:
This study involves conducting formative research to develop a culturally appropriate secondary prevention intervention for HIV-positive Black young men who have sex with men (B-YMSM). The intervention draws upon the principles of Critical Consciousness Theory (CCT). The formative research includes reviewing data and findings from relevant ATN protocols (i.e., 070, 068, and 073) and existing health promotion interventions targeting young men of color (i.e., the Young Warriors program, Hermanos de Luna y Sol [HLS]) and conducting focus groups with up to 32 HIV- positive B-YMSM.

DETAILED DESCRIPTION:
Focus groups will be conducted at two Adolescent Medicine Trials Unit (AMTU) sites and will guide the selection of the intervention content areas and the development of the intervention manual. The intervention aims to increase participation in health promoting behaviors and improve self-worth and self-concept among HIV-positive B-YMSM. Specifically, the intervention aims to address the following health promoting behaviors: 1) increasing engagement in HIV treatment; 2) improving medication adherence; 3) reducing sexual risk behaviors; 4) reducing substance use behaviors; and 5) increasing HIV status disclosure.

Based on reviews of ATN 070 data and existing related interventions (ATN 068, ATN 073, Young Warriors, HLS), draft components of the intervention curriculum for B-YMSM will be developed. Four focus groups will then be convened (two per AMTU) with HIV-positive B-YMSM to a) obtain input on the draft intervention curriculum, b) refine intervention components, and c) examine psychosocial factors that may mediate or moderate the intervention effect. The focus groups will be implemented using a "Rapid Approach" which allows for a focus on key areas of inquiry by asking fewer questions and focusing on targeted responses of focus group participants. All focus groups will be digitally recorded and transcribed. The transcripts will be reviewed and data analyzed using a phenomenological approach; protocol team members and members of two Youth Advisory Boards (YABs), which will include youth who are existing members of ATN site CABs as well as youth recruited from other local agencies and organizations), will work on the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

1. Receives services at one of the selected AMTU sites;
2. Male sex at birth and male gender at the time of the study;
3. Self identifies as "Black" (including Black/African-American, Black Latino, Black/Afro-Caribbean, Black/African immigrant, or any self-identified member of the African Diaspora);
4. HIV-infected as documented by medical record review or verification with referring medical professional;
5. Between the ages of 16-24 years inclusive at the time of consent;
6. HIV-infected through sexual behavior;
7. At least one sexual encounter involving oral or anal sex with a male partner in the past year;
8. Ability to understand both written and spoken English;
9. Willingness to participate in a focus group discussion with other HIV-positive B-YMSM; and
10. Willingness to provide signed informed consent or assent with parental permission as applicable for study participation.

Exclusion Criteria:

1. Active psychiatric condition that in the opinion of the site personnel would interfere with the ability to give true informed consent and to adhere to the study requirements;
2. Visibly distraught and/or visibly emotionally unstable (i.e., exhibiting suicidal, homicidal, or violent behavior);
3. Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with the ability to give true informed consent and to adhere to the study requirements;
4. Acute illness that, in the opinion of the treating clinician, would interfere with the participant's ability to adhere to the protocol requirements and/or interfere with the protocol objectives.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Produce an intervention focused on promoting critical consciousness among HIV-positive B-YMSM by using focus groups with HIV - positive B-YMSM | 1 year
  The focus groups will be conducted to:
  1. determine the needs of the intervention
  2. participants' views on the content areas that should and should not be included in the newly developed intervention
  3. participants' views on the following areas of intervention design will also be obtained:
     1. the critical consciousness coaching technique;
     2. program structure (e.g., frequency, length, time);
     3. format (group sessions, individual sessions, combined sessions, internet sessions, weekend retreats); (d) session content (e.g., prevention skills, content areas, study incentives).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wilson, PhD, Study Chair — Columbia University

REFERENCES:
- See also: ATN Website — https://www.atnonline.org